CLINICAL TRIAL: NCT02455115
Title: Renal Perfusion, Filtration and Oxygenation After Liver Transplantation -Effects of av Postoperative Blood Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Jenny Skytte Larsson, MD, Sahlgrenska University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MAP after Livertransplantation
Record Dates: First submitted 2015-04-23; First posted 2015-05-27 (Estimated); Last update posted 2016-09-28 (Estimated); Status verified 2016-09

CONDITIONS: Acute Kidney Injury; Liver Failure
Keywords: Acute kidney injury; Liver transplantation; Postoperative care; Glomerular filtration rate; Renal blood flow; Vasopressor; Norepinephrine
MeSH Terms: conditions — Acute Kidney Injury; Liver Failure | interventions — Norepinephrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 60 mmHg (Experimental): Alternating mean arterial pressure by lowering of the infusion rate of norepinephrine
  Interventions: Other: Alternating mean arterial pressure; Drug: Norepinephrine; Drug: Chromium ethylenediaminetetraacetic acid
- 75 mmHg (Experimental): Alternating mean arterial pressure by adjust of the infusion rate of norepinephrine
  Interventions: Other: Alternating mean arterial pressure; Drug: Norepinephrine; Drug: Chromium ethylenediaminetetraacetic acid
- 90 mmHg (Experimental): Alternating mean arterial pressure by augmentation of the infusion rate of norepinephrine
  Interventions: Other: Alternating mean arterial pressure; Drug: Norepinephrine; Drug: Chromium ethylenediaminetetraacetic acid

INTERVENTIONS:
Other: Alternating mean arterial pressure — In normovolemic patients directly after liver transplantation, target mean arterial pressure is altered using norepinephrine according to study protocol.
  Other Names: Norepinephrine
Drug: Norepinephrine — Infusion rate of norepinephrine is raised and lowered, respectively, in order to reach MAP 60, 75 and 90 mmHg in patients already requiring vasopressor for adequate blood pressure control.
  Other Names: Blood pressure control
Drug: Chromium ethylenediaminetetraacetic acid — Extraction of 51Cr-EDTA measured for FF and GFR
  Other Names: Infusion of 51Cr-EDTA

SUMMARY:
Comparing the effects of MAP 60, 75 and 90 mmHg, respectively, on renal blood flow, glomerular filtration rate and renal oxygen demand in patients with terminal liver failure directly after liver transplantation.

DETAILED DESCRIPTION:
Patients with terminal liver failure are at risk to develop postoperative acute kidney injury (AKI) after liver transplantation. This is associated with augmented morbidity (CRRT/HD), and mortality. Hypotension perioperatively is a risk factor for the development of postoperative AKI.

In the investigators' study, the researchers aim to investigate the importance of the level of mean arterial pressure (MAP) on functional renal parameters directly after liver transplantation. 12 patients will be included after given informed and written consent.

Directly after the operation, the patients stay sedated and ventilated, have reached normovolaemia and are in need of vasopressor for adequate blood pressure. MAP is varied using the vasopressor norepinephrine.

Central hemodynamics will be measured using arterial catheter, PiCCO and a central vein catheter.

Renal data measures (RBF (renal blood flow), RPF (renal plasma flow), FF (filtration fraction), GFR (glomerular filtration rate), RVR (renal vascular resistance), Arterial-renal vein oxygen content difference, RVO2 (renal oxygen consumption), and RO2extr (Renal oxygen extraction)), are conducted via a renal vein thermodilution catheter: A 8-Fr catheter is introduced into the left or right renal vein, via the right femoral vein under fluoroscopic guidance, position being confirmed by venography using ultra-low doses of iohexol.

After the collection of blood and urine blanks, an intravenous priming dose of chromium ethylenediaminetetraacetic acid (51Cr-EDTA) is given, followed by an infusion at a constant rate, individualized to BSA and preoperative serum creatinine. Serum 51Cr-EDTA activity from arterial and renal vein blood is measured using a well counter. FF is measured as extraction of Cr-EDTA.

After one hour and two control measurements and urine/blood sampling on baseline MAP 75 mmHg, the investigators will randomise to continue to MAP 90 mmHg or 60 mmHg reached by altering the infusion rate of norepinephrine. Measurements, blood sampling and urine collection according to the above description, are performed after 30 min at each level, finishing at 75 mmHg with two control measurements with 30 mins in between.

ELIGIBILITY:
Inclusion Criteria:

* Uncomplicated liver transplantation
* Age over 18 years
* Given informed consent preoperatively

Exclusion Criteria:

* Veno-venous bypass intraoperatively
* Uncontrolled postoperative bleeding
* Circulatory stability without need for vasopressor treatment
* Pronounced circulatory or respiratory instability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-01; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Change in Glomerular filtration rate (ml/min) | 60 min at baseline (75 mmHg), 30 min at randomized level 1(either 60 or 90 mmHg), 30 min at randomized level 2 (either 60 or 90 mmHg), 60 min after returning to baseline 75 mmHg again
  Change from baseline 75 mmHg to 60 and 90 mmHg, respectively

SECONDARY OUTCOMES:
Change in Renal blood flow (ml/min) | 60 min at baseline (75 mmHg), 30 min at randomized level 1(either 60 or 90 mmHg), 30 min at randomized level 2 (either 60 or 90 mmHg), 60 min after returning to baseline 75 mmHg again
  Measured via retrograde thermodilution catheter placed in renal vein. Change from baseline 75 mmHg to 60 and 90 mmHg, respectively.
Change in Renal oxygen consumption (ml/min) | 60 min at baseline (75 mmHg), 30 min at randomized level 1(either 60 or 90 mmHg), 30 min at randomized level 2 (either 60 or 90 mmHg), 60 min after returning to baseline 75 mmHg again
  Blood samples and measurements of blood flow via retrograde thermodilution catheter placed in renal vein.
  RBF × (CaO2-CrvO2) Change from baseline 75 mmHg to 60 and 90 mmHg, respectively
Change in Filtration fraction (%) | 60 min at baseline (75 mmHg), 30 min at randomized level 1(either 60 or 90 mmHg), 30 min at randomized level 2 (either 60 or 90 mmHg), 60 min after returning to baseline 75 mmHg again
  Extraction of Cr-EDTA, blood samples from renal vein catheter. Change from baseline 75 mmHg to 60 and 90 mmHg, respectively.
Change in Renal oxygen supply/demand relationship | 60 min at baseline (75 mmHg), 30 min at randomized level 1(either 60 or 90 mmHg), 30 min at randomized level 2 (either 60 or 90 mmHg), 60 min after returning to baseline 75 mmHg again
  Renal oxygen consumption compared to renal oxygen delivery (CaO2-CrvO2/CaO2). Change from baseline 75 mmHg to 60 and 90 mmHg, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Jenny Skytte Larsson, MD, Principal Investigator — Sahlgrenska University Hospital; Sven-Erik Ricksten, Professor, Study Chair — Sahlgrenska University Hospital
Locations (1):
- Sahlgrenska University Hospital, dpt of anesthesiology and intensive care, Gothenburg, VGR, Sweden

REFERENCES:
- [Derived] Skytte Larsson J, Bragadottir G, Redfors B, Ricksten SE. Renal function and oxygenation are impaired early after liver transplantation despite hyperdynamic systemic circulation. Crit Care. 2017 Apr 11;21(1):87. doi: 10.1186/s13054-017-1675-4. PMID 28395663